CLINICAL TRIAL: NCT05532982
Title: Barriers and Motivators Associated With Access to Care and Participation in Research Studies for Parkinson's Disease Among Asian Americans
Brief Title: Parkinson's Disease in Asian Americans
Status: Recruiting | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: Naheed Esar, Asian Women for Health (Unknown)
Responsible Party: Principal Investigator, Alice Tang, Professor, Tufts University
Other Study IDs: MJFF-020935
Record Dates: First submitted 2022-09-06; First posted 2022-09-08 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Parkinson's disease patients: Parkinson's disease patients of Asian descent
  Interventions: Other: Interviews and Surveys
- Parkinson's disease patients' care-givers: Care partners of Parkinson's Disease patients of Asian descent
  Interventions: Other: Interviews and Surveys
- Clinicians: Clinical providers of patients with Parkinson's disease, including physicians, nurses, nurse practitioners, physician assistants, physical therapists, etc.
  Interventions: Other: Interviews and Surveys
- Community stakeholders: Advocates for the Asian American community
  Interventions: Other: Interviews and Surveys

INTERVENTIONS:
Other: Interviews and Surveys — Qualitative interviews and surveys

SUMMARY:
The ultimate goal of this project is to use the findings to develop culturally appropriate programs and resources that can be disseminated to key stakeholders to improve access to PD care and increase inclusivity in PD research for Asian Americans. This study will serve as a first step towards developing broader community and patient education programs and active outreach campaigns to increase PD-specific literacy among Asian Americans. The results from this study will elucidate the role that language barriers, cultural perceptions, family influence, and other predisposing, enabling, or need factors have on delaying care for PD among Asian Americans. It will also provide much needed insight on how to improve inclusion of Asian Americans in PD research studies.

ELIGIBILITY:
Inclusion Criteria:

* Objective 1 (chart review):

  1. Chinese or Vietnamese ethnicity
  2. Age: 18 years of age or older
  3. Diagnosed or presented for PD care at the Tufts Medical Center (TMC) Movement Disorders Clinic (MDC) from January 1, 2010 to December 31, 2019.
* Objective 2 (qualitative study):

  1. Asian American person diagnosed with PD:

     1. Diagnosed with PD
     2. Chinese or Vietnamese ethnicity
     3. Age: 18 years of age or older
     4. Able to participate in an interview by phone or on Zoom
     5. Able to provide informed consent
  2. Primary caregivers of Asian American PD patients recruited into the study:

     1. Age: 18 years of age or older
     2. First-degree family member or spouse
     3. Self-identified as a primary caregiver of an Asian American person with PD
     4. Able to participate in an interview by phone or on Zoom
     5. Able to provide informed consent
  3. Clinicians:

     1. Any clinician (e.g. primary care provider, neurologist, resident, nurse, nurse practitioner, etc) that takes care of PD patients.
     2. Age: 18 years of age or older
  4. Key advocates in the Asian American community working specifically with the Asian elderly population.

     1. Employee or volunteer for a community-based organization working with the Asian elderly population (e.g. Greater Boston Chinese Golden Age Center, South Cove Manor, and Midtown Home Health Services) or other organizations working with PD patients and the elderly (e.g. Massachusetts Council on Aging and the Massachusetts Chapter of the American Parkinson's Disease Association)
     2. Age: 18 years of age or older
     3. Able to participate in a focus group discussion on Zoom

        Objective 3 (surveys of care partners of Asian American individuals with PD):

  <!-- -->

  1. Chinese or Vietnamese ethnicity
  2. Primary care partner of a family member with Parkinson's Disease
  3. Age: 18 years of age or older
  4. Care partner or family member with Parkinson's Disease must be of Asian descent

Exclusion Criteria:

Objective 1:

1. Patients diagnosed with juvenile-onset Parkinson's Disease

Objective 2:

PD patients only:

1. Patients with juvenile-onset Parkinson's Disease
2. Patients diagnosed with dementia
3. Patients on medication for cognitive impairment, e.g., anti-psychotics, donepezil (Aricept), rivastigmine (Exelon), and galantamine (Razadyne)

No exclusion criteria for other stakeholder groups (caregivers, clinical providers, key community advocates).

Objective 3:

1. Patients with juvenile-onset Parkinson's Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese and Vietnamese patients with Parkinson's disease and their care partners, clinicians, and community advocates.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Delay in seeking care | November 2022 - August 2024
  For the main outcome (delay in seeking care), the investigators will rely on self-report. Data obtained from Objectives 1 and 2 will be used to inform the development of a survey question (or a series of questions) that will capture this construct. The questionnaire will be piloted among a subgroup of participants recruited from the TMC MDC to calibrate the self-reported measure against data obtained from their medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided